CLINICAL TRIAL: NCT03483558
Title: Dietary Intervention Studies on a Variety of Vegetables
Brief Title: Vegetable Signature From Human Metabolomics Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Academia Sinica, Taiwan (Other); Tri-Service General Hospital (Other); Fu Jen Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NHRI_EC0991003
Record Dates: First submitted 2018-01-31; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-01

CONDITIONS: Vegetable Signature Documentation With Metabolomic Technique
Keywords: vegetable metabolite signature; human serum/urinary metabolite; liquid chromatography mass spectrometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Experimental): Participants were fed a standardized diet (without any vegetables) in this experiment.
  Interventions: Other: Control
- Spinach (Experimental): Participants were fed a standardized diet with 200g spinach in this experiment.
  Interventions: Other: Spinach
- Celery (Experimental): Participants were fed a standardized diet with 200g celery in this experiment.
  Interventions: Other: Celery
- Onion (Experimental): Participants were fed a standardized diet with 200g onion in this experiment.
  Interventions: Other: Onion
- Mixed Vegetables (Experimental): Participants were fed a standardized diet with 200g of mixed vegetables (spinach, celery, and onion) in this experiment.
  Interventions: Other: Mixed Vegetables

INTERVENTIONS:
Other: Control — A standardized diet without any vegetables was provided.
  Arms: Control
Other: Spinach — A standardized diet with 200g spinach was provided.
  Arms: Spinach
Other: Celery — A standardized diet with 200g celery was provided.
  Arms: Celery
Other: Onion — A standardized diet with 200g onion was provided.
  Arms: Onion
Other: Mixed Vegetables — A standardized diet with 200g of mixed vegetables (spinach, celery, and onion) was provided.
  Arms: Mixed Vegetables

SUMMARY:
The purpose of this study is to perform dietary intervention studies on a variety of vegetables.

DETAILED DESCRIPTION:
Plant-based foods have always been an important component of a healthy diet. High intake of plant foods may not only maintain normal bodily functions through the provision of dietary fiber, vitamins, and minerals but also relieve symptoms and prevent diseases. Many studies have pointed out that high intake of plant foods may reduce the incidence of non-communicable disease. Past research investigating the effect of phytochemicals has usually been limited to single substances or single foods. However, a number of researchers have pointed out that phytonutrients and dietary components are likely to act synergistically.Health effects and mechanisms of phytonutrients in combination have not been carefully studied in population settings. The technology of metabolomics has enabled the simultaneous measurement of hundreds of small molecules in biological samples. Exploring the change of metabolites after feeding can not only help us understand the role of plant foods, but may also provide opportunities to assess plant food intake levels.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5~30 kg/m2
* non-smoker
* non-alcoholic

Exclusion Criteria:

* Unwilling to stop taking the dietary supplements that may affect the experiment result.
* Unwilling to take the provided meal during the designated period.
* Taking hypertension or diabetes drugs.
* Diagnosed immune diseases (such as allergic diseases, autoimmune diseases, etc.), liver diseases, metabolic diseases (such as hyperthyroidism or hypothyroidism), or other not suitable for the dietary study.
* Diagnosed cancer or other severe diseases.
* Suffered from urinary tract infection or took antibiotic in the past three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06-11 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2015-05-28 (Actual)

PRIMARY OUTCOMES:
Intensities of multiple serum metabolites | Baseline (fasting state before breakfast at 7:30AM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 4 Hours (immediately before lunch at 11:30AM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 5.5 hours (after lunch at 13:00PM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 6.5 hours (after lunch at 14:00 PM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 7.5 hours (after lunch at 15:00PM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 8.5 hours (after lunch at 16:00PM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 9.5 hours (after lunch at 17:00PM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 10.5 hours (after lunch at 18:00PM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple serum metabolites | 11.5 hours (after lunch at 19:00PM)
  The outcome measure consists of intensities of multiple serum metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple urinary metabolites | Baseline (overnight urine sample collected at 7:30AM)
  The outcome measure consists of intensities of multiple urinary metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple urinary metabolites | 3.5~4 hours (before lunch urine sample collected during 11:00~11:30AM)
  The outcome measure consists of intensities of multiple urinary metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple urinary metabolites | 4.5~6.5 hours (2-hour after lunch urine sample collected from 12:00 to 14:00PM)
  The outcome measure consists of intensities of multiple urinary metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple urinary metabolites | 6.5~8.5 hours (4-hour after lunch urine sample collected from 14:00 to 16:00PM)
  The outcome measure consists of intensities of multiple urinary metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.
Intensities of multiple urinary metabolites | 8.5~11.5 hours (7-hour after lunch urine sample collected from 16:00 to 19:00PM)
  The outcome measure consists of intensities of multiple urinary metabolites from a liquid chromatography/time-of-flight/mass spectrometry (LC/TOF/MS) experiment. Intensity means the level of response variable (a given metabolite) showing the degree of response detected by LC/TOF/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — National Health Research Institutes, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided